CLINICAL TRIAL: NCT05246137
Title: A Phase III, Open Label, Single Arm, Multi-centre, Trial to Assess the Safety and Immunogenicity of a Booster Vaccination With a Recombinant Protein RBD Fusion Heterodimer Candidate (PHH-1V) Against SARS-CoV-2, in Adults Vaccinated Against COVID-19.
Brief Title: A Phase III Trial to Assess the Safety and Immunogenicity of a HIPRA's Candidate Booster Vaccination Against COVID-19.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hipra Scientific, S.L.U (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HIPRA-HH-5
Record Dates: First submitted 2022-02-08; First posted 2022-02-18 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; SARS-CoV-2 Acute Respiratory Disease
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: COVID-19 Vaccine HIPRA 40 ug/dose (Experimental): COVID-19 Vaccine HIPRA, where subjects will receive one intramuscular injection of COVID-19 vaccine developed by HIPRA
  Interventions: Biological: COVID-19 Vaccine 40 ug/dose

INTERVENTIONS:
Biological: COVID-19 Vaccine 40 ug/dose — Intramuscular injection of 0,5 ml with 40 ug of recombinant PHH-1V

SUMMARY:
This is a phase III clinical study to assess the safety, tolerability and immunogenicity of PHH-1V as a booster dose in healthy adult subjects vaccinated against COVID-19 with the Comirnaty, Spikevax, Vaxevria or Janssen vaccine.

DETAILED DESCRIPTION:
This is a phase III clinical study to assess the safety, tolerability and immunogenicity of PHH-1V as a booster dose in healthy adults vaccinated against COVID-19 with the Comirnaty, Spikevax, Vaxevria or Janssen vaccine at least 91 days before day 0. All the participants will receive a booster dose of the HIPRA's COVID-19 Vaccine and will be followed for 26 weeks or 52 weeks if they participate in the safety cohort, or the immunogenicity cohort, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥ 16 years old at Day 0.
* Willing to provide consent indicating that she or he understands the purpose and potential risks and is willing and able to participate in the study and comply with all the study requirements and procedures.
* Have a recognized primary vaccination scheme recognized by the authorities with Comirnaty, Spikevax, Vaxevria or Janssen at least 91 days and preferably a maximum of 240 days before Day 0.
* If having an underlying illnesses must be stable and well-controlled according to the investigator judgment.
* Participant is willing to avoid receiving live attenuated vaccines (licensed) within 4 weeks before screening or after receiving any study vaccine, or other not live vaccines (licensed) within 14 days before and after receiving any study vaccine.
* Participant agrees not to donate blood, blood products and bone marrow at least 3 months before and after vaccination.
* Female participant of childbearing potential must have a negative pregnancy test on the on Day 0 prior to vaccination.
* Female participant of childbearing potential must use any acceptable contraceptive method that should be started on day 0 and until 8 weeks after vaccination (hormonal contraception: oral, injectable or transdermal patch, intrauterine device, vasectomized partner, sexual abstinence or condom).
* Male participants must use any acceptable contraceptive method that should be started on day 0 and until 8 weeks after vaccination (vasectomized participants, condom, sexual abstinence).
* Male participants must refrain from donating sperm for at least 28 days after day 0.

Exclusion Criteria:

* History of anaphylaxis to any prior vaccine.
* Previous severe SARS-CoV-2 infections that required >24 hous of hospitalisation.
* Participant received or plans to receive live attenuated vaccines within 4 weeks before and after day 0; or other not live vaccines within 14 days before and after day 0.
* Pregnancy or breast-feeding at screening or Day 0 or willingness/intention to become pregnant during the study.
* Having a clinically significant acute illness or fever (temperature ≥38º C (100.4ºF)) at screening or within 48 hours prior to Day 0.
* Participant had a surgery requiring hospitalization before vaccination and he/she has not received the hospital discharge at day 0; or has a surgery requiring hospitalization planned within 12 weeks after study vaccine administration.
* Having any active malignancy even if under treatment except for non-melanoma skin cancer, uterine cervical carcinoma, anal carcinoma, localized prostate cancer.
* Having ongoing severe and non-stable psychiatric condition likely to affect participation in the study.
* Having problematic or risk use of substances including alcohol that can compromise the study follow-up.
* Having a bleeding disorder or has any condition that in the opinion of the investigator contraindicates intramuscular injections.
* Having abnormal function of the immune system, except stable clinical conditions like controlled HIV.
* Having clinically significant and unstable cardiovascular, respiratory, hepatic, neurological, gastrointestinal, renal, or any other medical disorder judged by the investigator within 3 months before screening.
* Chronic or recurrent administration of systemic immunosuppressant medication.
* Having received immunoglobulins and/or blood-derived products 12 weeks prior vaccination (Day 0) or expects to receive them during the study.
* Having received any immunotherapy (monoclonal antibodies, plasma) aimed to prevent or treat COVID-19 within 90 days before day 0.
* Participation in any research involving an investigational product (drug, biologic, device) within 12 weeks prior to vaccination and during the study.
* Participant has donated ≥ 450ml of blood products within 12 weeks before screening.
* Participant has any medical condition and/or finding that in the investigator opinion might increase participant risks, interfere with the study or impair interpretation of study data.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2646 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and tolerability) | Day 7
  Number, percentage, and characteristics of solicited local and systemic reactions through Day 7 after vaccination.
Incidence of Treatment-Emergent Adverse Events (Safety and tolerability) (AEs) | Day 28
  Number, percentage, and characteristics of unsolicited local and systemic adverse events (AEs) through Day 28 after vaccination
Incidence of Serious Adverse Events (Safety and tolerability) (SAE) | Day 365
  Number and percentage of serious adverse events (SAEs) through the end of the study.
Incidence of Special Interest Adverse Events (Safety and tolerability) (AESI). | Day 365
  Number and percentage of adverse event of special interest (AESI) through the end of the study.
Incidence of Medically Attended Adverse Events (Safety and tolerability) (MAAEs) | Day 365
  Number and percentage of medically attended adverse events (MAAE) related to study vaccine through the end of the study.
Incidence of Adverse Events in laboratory parameters (Safety and tolerability) | Day 365
  Grade 3 and 4 changes from baseline in safety laboratory parameters at Days 14, 91 and 182 after vaccination.
  through the end of the study.

SECONDARY OUTCOMES:
Changes in the immunogenicity measured by pseudovirus neutralisation | Day 365
  Neutralisation titre against Wuhan and Omicron strains, and any other relevant VOC in the epidemiologic moment, measured as inhibitory concentration 50 (IC50) by a pseudovirion-based neutralisation assay (PBNA) and reported as reciprocal concentration for each individual sample and geometric mean titre (GMT) for descriptive statistics analysis at Baseline and at Days 14, 91, 182 and 365.
Changes in the immunogenicity measured by pseudovirus neutralisation | Day 14
  The geometric mean fold rise (GMFR) in neutralising antibody titre from baseline to Day 14.
Changes in the immunogenicity measured by means of total antibody against RBD | Day 365
  Binding antibodies titre measured for each individual sample and GMT for descriptive statistics analysis at Baseline and Days 14, 91, 182 and 365.
Changes in the immunogenicity measured by means of total antibody against RBD. | Day 14
  The geometric mean fold rise (GMFR) in binding antibody titre from baseline to Day 14.
Changes in the immunogenicity measured by means of total antibody against RBD | Day 14
  The percentage of subjects that after the booster dose have a ≥4-fold change in binding antibodies titre from Baseline to Day 14.

OTHER OUTCOMES:
To assess number of subjects with SARS-CoV-2 infections ≥14 days after PHH-1V booster. | Day 365
  Number and percentage of subjects with SARS-CoV-2 infections ≥14 days after PHH-1V booster according to COVID-19 infection criteria throughout the study duration.
To assess number of COVID-19 severe infections ≥14 days after receiving PHH-1V. SARS-CoV-2 infections ≥14 days after PHH-1V booster. | Day 365
  Number and percentage of COVID-19 severe infections ≥14 days after PHH-1V booster and through the end of the study.
To assess number of COVID-19 severe infections ≥14 days after receiving PHH-1V and hospital admissions SARS-CoV-2 infections ≥14 days after PHH-1V booster. | Day 365
  Number and percentage of hospital admissions associated with COVID-19 ≥14 days after PHH-1V booster and through the end of the study.
To assess number of COVID-19 severe infections ≥14 days after receiving PHH-1V in ICU. SARS-CoV-2 infections ≥14 days after PHH-1V booster. | Day 365
  Number and percentage of intensive care unit (ICU) admissions associated with COVID-19 ≥14 days after PHH-1V booster and through the end of the study.
To assess number of COVID-19 severe infections ≥14 days after receiving PHH-1V receiving noninvasive ventilation. SARS-CoV-2 infections ≥14 days after PHH-1V booster. | Day 365
  Number and percentage of noninvasive ventilation administration associated with COVID-19 ≥14 days after PHH-1V booster and through the end of the study.
To assess number of COVID-19 severe infections ≥14 days after receiving PHH-1V causing death. | Day 365
  Number and percentage of deaths associated with COVID-19 ≥14 days after PHH-1V booster and through the end of the study.
To evaluate T-cell mediated responses against the SARS-CoV-2 S glycoprotein at Baseline and Day 14 in subjects who have received two doses of Vaxzevria vaccine and PHH-1V as a booster.. | Day 14
  T-cell-mediated response to the SARS-CoV-2 S protein as measured by whole peripheral blood mononuclear cell (PBMC) stimulation by enzyme-linked immune absorbent spot (ELISpot) at Baseline and at Day 14. This analysis will be performed in 30 subjects.
To assess Th-1/Th-2 T-cell mediated responses against S protein at Baseline and Day 14 in subjects who have received two doses of Vaxzevria vaccine and PHH-1V as a booster. | Day 14
  CD4+/CD8+ T-cell response to the SARS-CoV-2 S protein as measured by in vitro PBMC stimulation by cytokine staining assays at Baseline and at Day 14. This analysis will be performed in 30 subjects.

CONTACTS AND LOCATIONS:
Locations (18):
- Hospital de Niguarda, Milan, Italy
- Spain (17):
  - Hospital Germans Trias I Pujol, Badalona, Barcelona
  - Hospital de Mollet, Mollet del Vallès, Barcelona
  - Hospital Principe de Asturias, Meco, Madrid
  - Hospital HM Puerta del Sur, Móstoles, Madrid
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital HM Delfos, Barcelona
  - Hospital Quironsalud Barcelona, Barcelona
  - Hospital Vall Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Dr. Josep Trueta, Girona
  - Hospital Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital HM Sanchinarro, Madrid
  - Hospital Quironsalud Madrid, Madrid
  - Hospital HM Montepríncipe, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Clínico de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moros A, Prenafeta A, Barreiro A, Perozo E, Fernandez A, Canete M, Gonzalez L, Garriga C, Pradenas E, Marfil S, Blanco J, Cebollada Rica P, Sistere-Oro M, Meyerhans A, Prat Cabanas T, March R, Ferrer L. Immunogenicity and safety in pigs of PHH-1V, a SARS-CoV-2 RBD fusion heterodimer vaccine candidate. Vaccine. 2023 Aug 7;41(35):5072-5078. doi: 10.1016/j.vaccine.2023.07.008. Epub 2023 Jul 16. PMID 37460353